CLINICAL TRIAL: NCT05585606
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter Study of the Safety and Neuroprotective Capacity of Scp776 in Subjects Undergoing Endovascular Thrombectomy for Acute Ischemic Stroke
Brief Title: Study of the Safety and Neuroprotective Capacity of Scp776 in Acute Ischemic Stroke
Acronym: ARPEGGIO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Silver Creek Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SCP-CL-0003
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke (AIS)
Keywords: Stroke, Acute; Neuroprotectant
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: This is a Phase 2 randomized, placebo-controlled, double-blind study that will be conducted in 2 parts: sequential dose escalation in Part A, followed by dose expansion in Part B.
  In Part A, approximately 60 evaluable subjects will be assigned 1:1:1:3 overall to Cohort 1, Cohort 2, Cohort3, or placebo.
  Doses of scp776 will be tested sequentially in 3 cohorts, each in parallel with a volume-matched placebo randomized as 1:1 scp776:placebo within each cohort, to maintain the overall 1:1:1:3 ratio.
  Subjects will receive doses of either normal saline (placebo) or scp776, approximately 24 hours apart.
  * Cohort 1 dose regimen:
    - 1.9 mg/kg
  * Cohort 2 dose regimen:
    - 3.8 mg/kg
  * Cohort 3 dose regimen:
    * 4.8 mg/kg
  The study will proceed into Part B (dose expansion), in which approximately 40 subjects will be randomized 3:1 to the chosen scp776 therapeutic dose from Part A or volume-matched placebo:
  Cohort 3: Therapeutic dose scp776:placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Volume Matched Placebo (normal saline)
  Interventions: Drug: Placebo
- scp776 (1.9 mg/kg) (Experimental): Cohort 1 dose regimen:
  Intravenous (IV) injection(s) over 2 minutes
  - 1.9 mg/kg
  Interventions: Drug: scp776 (1.9 mg/kg); Drug: scp776 (all dose levels)
- scp776 (3.8 mg/kg) (Experimental): Cohort 2 dose regimen:
  Intravenous (IV) injection(s) over 2 minutes
  - 3.8 mg/kg
  Interventions: Drug: scp776 (3.8 mg/kg); Drug: scp776 (all dose levels)
- scp776 (4.8 mg/kg) (Experimental): Cohort 3 dose regimen: Intravenous (IV) injection(s) over 2 minutes - 4.8 mg/kg
  Interventions: Drug: scp776 (4.8 mg/kg); Drug: scp776 (all dose levels)

INTERVENTIONS:
Drug: Placebo — Volume Matched Placebo
  Arms: Placebo
Drug: scp776 (1.9 mg/kg) — Cohort 1 dose regimen:
  Intravenous (IV) slow injection(s) over 2 minutes
  - 1.9 mg/kg
  Arms: scp776 (1.9 mg/kg)
Drug: scp776 (3.8 mg/kg) — Cohort 2 dose regimen:
  Intravenous (IV) slow injection(s) over 2 minutes
  - 3.8 mg/kg
  Arms: scp776 (3.8 mg/kg)
Drug: scp776 (4.8 mg/kg) — Cohort 3 dose regimen: Intravenous (IV) slow injection(s) over 2 minutes - 4.8 mg/kg
  Arms: scp776 (4.8 mg/kg)
Drug: scp776 (all dose levels) — A composite group encompassing all participants who received any dose level of the investigational drug under evaluation.
  Arms: scp776 (1.9 mg/kg); scp776 (3.8 mg/kg); scp776 (4.8 mg/kg)

SUMMARY:
A Randomized, Placebo-Controlled, Double-Blind, Multicenter Study of the Safety and Neuroprotective Capacity of Scp776 in Subjects Undergoing Endovascular Thrombectomy for Acute Ischemic Stroke

DETAILED DESCRIPTION:
This is a Phase 2 randomized, placebo-controlled, double-blind study that will be conducted in 2 parts: sequential dose escalation in Part A, followed by dose expansion in Part B.

In Part A, approximately 60 evaluable subjects will be assigned 1:1:1:3 overall to Cohort 1, Cohort 2, Cohort 3, or placebo. Doses of scp776 will be tested sequentially in 3 cohorts, each in parallel with a volume-matched placebo randomized as 1:1 scp776:placebo within each cohort, to maintain the overall 1:1:1:3 ratio.

Subjects will receive doses of either normal saline (placebo) or scp776, approximately 24 hours apart.• Cohort 1 dose regimen:- 1.9 mg/kg• Cohort 2 dose regimen:- 3.8 mg/kg• Cohort 3 dose regimen:- 4.8 mg/kg

Upon completion of Part A, the study will proceed into Part B (dose expansion), in which approximately 40 subjects will be randomized 3:1 to the chosen scp776 therapeutic dose from Part A or volume-matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Body weight of less than 150 kg.
* AIS intended for immediate endovascular treatment.
* Disabling stroke defined as a baseline NIHSS ≥6 at the time of randomization.
* Confirmed symptomatic intracranial occlusion, based on qualifying imaging, at one or more of the following locations: intracranial carotid artery and/or M1 or M2 middle cerebral artery.
* Onset of AIS (last time subject seen well) to randomization is ≤24 hours.
* Intended endovascular treatment with an approved endovascular device.
* Pre-AIS (24 hours before stroke onset) independent functional status in activities of daily living with Modified Rankin Scale score of 0, 1, or 2. Subject must be living in their own home, apartment, or seniors' lodge where no nursing care is required.
* Treating team and subject family are committed to full medical support for the subject.
* Signed informed consent from subject or legally authorized representative, if required to enable inclusion by applicable national laws and regulations and the applicable independent review boards/ethics committee requirements for obtaining consent. Electronic consent is allowed in jurisdictions wherein this consent process is allowed.
* Biologically female subjects must meet the following:

  1. Subject must be surgically sterile or be at least 1 year postmenopausal, OR
  2. Subjects of child-bearing potential must:

  i. have a negative serum or urine pregnancy test at Screening, AND ii. have no plans to become pregnant or to breast feed during the study, AND iii. at least one of the following must apply:
  1. have a monogamous partner who is surgically sterile.
  2. have a monogamous same sex partner.
  3. be practicing abstinence or using an acceptable form of birth control while participating in the study through Day 90. Site personnel will provide instructions on what is an acceptable method.
* If male, unless the subject has a same sex partner, be either sterile (surgically or biologically), commit to an acceptable double barrier method of birth control, or practice abstinence, until at least 30 days after study drug administration. Site personnel will provide instructions on what is an acceptable method.

Exclusion Criteria:

* Evidence of acute intra-cerebral hemorrhage on qualifying imaging, per radiology lab manual.
* Poor/no collateral circulation in the opinion of the investigator (e.g., collateral score of 0 or 1 if data available).
* ASPECT score of 0-4.
* Current AIS is being treated with IV thrombolytic therapy (e.g., alteplase, tenecteplase), or the subject has received thrombolytic therapy within the previous 24 hours.
* Intent to use any endovascular device that is not Food and Drug Administration (FDA)-approved.
* Planned use of intra arterial thrombolytic therapy.
* Known severe contrast allergy or absolute contraindication to iodinated contrast preventing endovascular intervention.
* Clinical history, past imaging, or clinical judgment suggests that the intracranial occlusion is chronic or there is suspected intracranial dissection such that there is a predicted lack of success with endovascular intervention.
* Known arterial condition that would prevent the mechanical device from achieving reperfusion (e.g., aortic dissection, carotid stent).
* Subjects with end stage kidney disease.
* Part A Cohort 1: Subjects taking a chronic anticoagulant (e.g., apixaban, warfarin) are excluded. Chronic use of anti-platelet drugs is acceptable.
* Part A Cohort 2: Subjects taking a chronic anticoagulant (e.g., apixaban, warfarin) are excluded unless subject has both a STAT international normalized ratio (INR) < 1.7, and a platelet count > 100K/µL prior to randomization. Chronic use of anti-platelet drugs is acceptable.
* Part A Cohort 3 and Part B: With SRC approval, subjects in Part A Cohort 3 and Part B taking a chronic anticoagulant (e.g., apixaban, warfarin) are excluded unless subject has both a STAT international normalized ratio (INR) < 1.7, and a platelet count > 100K/µL prior to randomization.

(If the SRC does not approve expansion of this criterion, then subjects taking a chronic anticoagulant (e.g., apixaban, warfarin) are excluded, as in Cohort 1. Chronic use of anti-platelet drugs is acceptable in either case.)

* Known metastatic malignancy with poor prognosis.
* Subjects with any comorbid disease, condition, or situation that would confound the neurologic and functional evaluations, prevent improvement, or render the subject unable to complete follow-up treatment, in the opinion of the investigator. Examples of excluded comorbid conditions include respiratory failure because of pneumonia, chronic diseases with significant disability, or non-ambulatory status. Contact medical monitor for consultation if necessary.
* Participation in another clinical trial of an FDA-unapproved therapeutic device or drug in the 30 days preceding study inclusion.
* Subject was a participant in either SCP CL 0001 or SCP CL 0002 and received scp776, or previously participated in SCP-CL-0003.
* Subject is experiencing moderate or severe hypotension as defined by CTCAE criteria (i.e., symptomatic and requiring medical intervention with fluid resuscitation and/or vasopressors) or a confirmed systolic blood pressure less than 90 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Total number of SAEs recorded prior to hospital discharge | Baseline to Day 7 or at hospital discharge (whichever occurs first).
  Generalized linear models will be fit assuming a Poisson family with log link. The regression model will include a term for the duration of hospitalization. The regression models may also be adjusted for any or all of the following utilizing a stepwise approach: Time from LKW or stroke onset to reperfusion; Reperfusion Status (eTICI score from central read); Age; and, ASPECTS (raw score from central read).
Proportion of subjects experiencing adverse events of special interest (AESIs) | Baseline to Day 7 or at hospital discharge (whichever occurs first).
  Proportion of subjects experiencing adverse events of special interest (AESIs):
  * Hypoglycemia
  * Tachycardia
  * Bleeding events:
    * Symptomatic intracranial hemorrhage as per the central imaging review
    * Asymptomatic intracranial hemorrhage as per the central imaging review
    * Extracranial hemorrhage

SECONDARY OUTCOMES:
NIH Stroke Scale (NIHSS) Score at Day 7 / Discharge (whichever comes first) | Baseline to Day 7 or at hospital discharge (whichever occurs first).
  NIH Stroke Scale score assessing neurological deficits and stroke severity. Scores range from 0 (no deficits) to 42 (severe deficits).
  NIHSS at discharge will be analyzed using Analysis of Covariance (ANCOVA). Terms to be included in the model are age, baseline NIHSS, ASPECTS, reperfusion status (TICI-based reperfusion grade), and treatment.
NIH Stroke Scale (NIHSS) Score | Daily from Days 1 through 7, Day 30, and Day 90.
  NIH Stroke Scale (NIHSS) score assessing neurological deficits and stroke severity. Scores range from 0 (no deficits) to 42 (severe deficits).
Modified Rankin Scale (mRS) Score | Day 7 or discharge (whichever occurs first), Day 30, and Day 90.
  Assessment of disability after stroke using the Modified Rankin Scale, ranging from 0 (no disability) to 6 (death).
Infarct Volume by Central Imaging Review | At 24 hours, and 72 - 96 hours or discharge (whichever occurs first).
  Infarct volume measured centrally via imaging (MRI or CT), evaluating ischemic lesion size.
All-cause Mortality | By Day 30, and by Day 90.
  Incidence of death from any cause.

OTHER OUTCOMES:
Duration of Hospitalization | Baseline to Day 90 or at hospital discharge (whichever occurs first).
  Number of consecutive days of inpatient hospitalization following the qualifying acute ischemic stroke.
Barthel Index Score at Day 90 | Day 90.
  Assessment of functional independence in activities of daily living (ADL). Scores range from 0 (complete dependence) to 100 (complete independence).
Proportion of Patients Achieving Barthel Index Score ≥90 | Day 90.
  Percentage of patients achieving Barthel Index scores of 90-100, indicating minimal or no dependence in daily living activities.
Exploratory Pharmacodynamics (PD) of Scp776 in this Population | Multiple post-dose timepoints up to 72 hours.
  Evaluation of exploratory pharmacodynamic effect via blood glucose area under the concentration-time curve (glucose AUC).
Area Under the Concentration-Time Curve of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - area under the concentration time curve from time 0 to the last observed non-zero concentration (AUC0-t).
Extrapolated Area Under the Concentration-Time Curve of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-inf).
Serum Concentration at End of Injection of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - serum drug concentration at the end of injection (Ceoi).
Volume of Distribution of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - apparent volume of distribution during the terminal elimination phase (Vz).
Total Serum Clearance of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - apparent total serum clearance after intravenous (IV) administration (CL).
Elimination Rate Constant of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - apparent first order terminal elimination rate constant (Kel).
Elimination Half-Life of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - apparent first order terminal elimination half-life (t½).
Maximum Observed Concentration of Scp776 | Pre-dose and multiple post-dose timepoints up to Day 30.
  Pharmacokinetic parameter assessed using noncompartmental methods following intravenous administration of scp776 - Maximum observed concentration (Cmax).
Immunogenicity Evaluation of Scp776 | Pre-dose and multiple post-dose timepoints up to study completion (approximately Day 90).
  Evaluation of anti-drug antibody (ADA) formation in response to scp776 treatment. Presence of ADA measured at specified timepoints.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Banner University Medical Center /Univ of Arizona, Tucson, Arizona
  - Hartford Hospital, Hartford, Connecticut
  - Marcus Neuroscience Institute, Boca Raton, Florida
  - University of Miami - Jackson Memorial Hospital, Miami, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - SSM Health DePaul Hospital, Bridgeton, Missouri
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - UNM Hospital, Albuquerque, New Mexico
  - Northshore University Hospital, Manhasset, New York
  - Lennox Hill Hospital, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Mercy Health - St Vincent Medical Center, Toledo, Ohio
  - Mercy Health - St Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Stroke Center at OHSU, Portland, Oregon
  - Providence St. Vincent Medical Center, West Haven-Sylvan, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Penn State Health - M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - Medical College of Wisconsin and Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No